CLINICAL TRIAL: NCT06504290
Title: A Phase I Clinical Study Evaluating the Safety, Tolerability, and Pharmacokinetics of VV119 Capsules With Multiple Ascending Doses in Chinese Healthy Adult Subjects and Patients With Schizophrenia
Brief Title: Evaluating Safety, Tolerability and Pharmacokinetic of Multiple Ascending Doses of VV119
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vigonvita Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VV119-02
Record Dates: First submitted 2024-07-02; First posted 2024-07-16 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part Ⅰ- in healthy adult subjects (Experimental)
  Interventions: Drug: VV119 Placebo （in healthy adult subjects）; Drug: VV119 （in healthy adult subjects）
- Part Ⅱ-in adult patients with schizophrenia (Experimental)
  Interventions: Drug: VV119(in adult patients with schizophrenia); Drug: VV119 Placebo （in adult patients with schizophrenia）

INTERVENTIONS:
Drug: VV119 Placebo （in healthy adult subjects） — VV119 0.5 mg Group:2 subjects will receive VV119 Placebo 0.5 mg, orally once daily for 14 days.
  VV119 1 mg Group:2 subjects will receive VV119 Placebo 1 mg, orally once daily for 14 days.
  Arms: Part Ⅰ- in healthy adult subjects
Drug: VV119 （in healthy adult subjects） — VV119 0.5 mg Group:6 subjects will receive VV119 0.5 mg, orally once daily for 14 days.
  VV119 1 mg Group:6 subjects will receive VV119 1 mg, orally once daily for 14 days.
  Arms: Part Ⅰ- in healthy adult subjects
Drug: VV119(in adult patients with schizophrenia) — VV119 2 mg Group:6 subjects will receive 2 0.5mgVV119 capsules on the first four days, then take 1 2mgVV119 capsules and 1 0.5mg VV119 Placebo from the fifth day to the 28th day， orally once daily, VV119 4 mg Group:6 subjects will receive 2 0.5mgVV119 capsules on the first four days, take 1 2mgVV119 capsules and 1 0.5mg VV119 Placebo from the fifth day to the seventh day , then 2 2mgVV119 capsules and 1 0.5mg VV119 Placebo from the eighth day to the 28th day ,orally once daily, VV119 6 mg Group:6 subjects will receive 2 0.5mgVV119 capsules on the first three days,take 1 2mgVV119 capsules and 1 0.5mg VV119 Placebo from the forth day to the fifth day , take 2 2mgVV119 capsules and 1 0.5mg VV119 Placebo from the sixth day to the seventh day , then 3 2mgVV119 capsules and 1 0.5mg VV119 Placebo from the eighth day to the 28th day ,orally once daily.
  Arms: Part Ⅱ-in adult patients with schizophrenia
Drug: VV119 Placebo （in adult patients with schizophrenia） — VV119 2 mg Group:2 subjects will receive 1 0.5mgVV119 capsules and 1 0.5mg VV119 Placebo on the first four days, then take 1 2mgVV119 Placebo and 1 0.5mg VV119 capsules from the fifth day to the 28th day， orally once daily, VV119 4 mg Group:2 subjects will receive 1 0.5mgVV119 capsules and 1 0.5mg VV119 Placebo on the first four days, take 1 2mgVV119 Placebo and 1 0.5mg VV119 capsules from the fifth day to the seventh day , then 2 2mgVV119 Placebo and 1 0.5mg VV119 capsules from the eighth day to the 28th day ,orally once daily, VV119 6 mg Group:2 subjects will receive 1 0.5mgVV119 capsules and 1 0.5mg VV119 Placebo on the first three days, take 1 2mgVV119 Placebo and 1 0.5mg VV119 capsules from the forth day to the fifth day ,take 2 2mgVV119 capsules and 1 0.5mg VV119 Placebo from the sixth day to the seventh day, then 3 2mgVV119 Placebo and 1 0.5mg VV119 capsules from the eighth day to the 28th day ,orally once daily.
  Arms: Part Ⅱ-in adult patients with schizophrenia

SUMMARY:
This study will consist of 2 parts: Part Ⅰ-in healthy adult subjects, Part Ⅱ-in adult patients with schizophrenia

DETAILED DESCRIPTION:
Part Ⅰ was designed as single-center, randomized, double-blind, placebo-controlled, dose-escalation trial to assess the safety, tolerability, pharmacokinetics （PK） of multiple doses of VV119 in Chinese healthy adult subjects.

Part Ⅱ was designed as multicenter, randomized, double-blind, placebo-controlled, dose-escalation trial to assess the safety, tolerability, pharmacokinetics （PK） and efficacy of multiple doses of VV119 in adult patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

Healthy adult subjects：

1. Males: aged 18 to 45 years old, Body weight no less than 50.0kg; females: Aged 18 to 60 years old, Body weight no less than 45.0kg, Body Mass Index of 19.0 to 26.0kg/m2.
2. Medically healthy, physical examination, vital signs examination, laboratory examination, electrocardiogram examination results were normal or abnormal without clinical significance.
3. Males' subjects who are willing to take effective contraceptive during the study and within 6 months after the study completed; females of non-child-bearing potential.
4. Subjects who are able to understand and follow study plans and instructions; Subjects who have voluntarily decided to participate in this study and signed the informed consent form.

Adult patients with schizophrenia:

1. Aged 18 to 65 years old, Body Mass Index of 18.5 to 30kg/m2, males, Body weight no less than 50.0kg; females: Body weight no less than 45.0kg.
2. Males' subjects who are willing to take effective contraceptive during the study and within 6 months after the study completed; females of non-child-bearing potential.
3. Subject has a primary diagnosis of schizophrenia established by a comprehensive psychiatric evaluation based on the DSM-5 and MINI at least 1 year.
4. Subject is experiencing an acute exacerbation or relapse of psychotic symptoms.
5. PANSS total score at least 70 and CGI-S score of ≥4 at screening.
6. Subjects who have a history of antipsychotics.
7. The subjects and their guardians fully understand the purpose and requirements of the trial, voluntarily participate in the clinical trial and sign the written informed consent form and are willing to complete the whole trial process according to the trial requirements.

Exclusion Criteria:

Healthy adult subjects：

1. With current or past medical history diseases or dysfunction that affect the clinical trial, evaluated by the investigator, including but not limited to central nervous system, cardiovascular system, respiratory system, digestive system, urinary system, endocrine system, blood system, ophthalmology and other diseases, history of malignant tumor or other diseases that are not suitable for participating in the clinical trial.
2. With current or previous mental disorders and brain dysfunction, or suicide risk according to the clinical judgment of the investigator, or a history of self-mutilation.
3. With any surgical condition or condition that may significantly affect the absorption, distribution, metabolism and excretion of the drug, or may pose a hazard to the subjects participating in the trial, such as history of gastrointestinal surgery (gastrectomy, gastrointestinal anastomosis, intestinal resection, etc.), urinary tract obstruction or dysuria, gastroenteritis, gastrointestinal ulcers, history of gastrointestinal bleeding, etc.
4. With a known history of allergy to investigating drug ingredients or similar drugs, a history of allergic diseases or allergic constitution.
5. Positive for hepatitis B virus surface antigen （HBsAg）, or syphilis antibody (Anti-TP), or hepatitis C antibody (anti-HCV), or human immunodeficiency virus antigen/antibody combined detection (HIV-Ag/Ab).
6. With a history of surgery within 3 months before screening, or have not recovered from surgery, or have an expected surgical plan during the trial.
7. With a blood donation or blood loss ≥ 400mL within 3 months before screening, or a blood donation or blood loss ≥ 200mL within 1 month, or a history of blood product use within 3 months before screening.
8. Taking any prescription drugs, over-the-counter drugs, and any functional vitamins or herbal products within 2 weeks before screening.
9. Using any drugs that inhibit or induce hepatic drug metabolizing enzymes CYP3A4, CYP3A5, CYP2D6 (such as inducers - phenobarbital, rifampicin, carbamazepine, phenytoin sodium, glucocorticoids, etc.; inhibitors - ketoconazole, itraconazole, cimetidine, clarithromycin, verapamil, erythromycin, etc.) within 4 weeks (or 5 half-lives, whichever is longer) before screening.
10. Participating in any clinical trial and taking clinical trial drugs within 3 months before screening, or being participating in other clinical trials.
11. Smoke test positive or smoking more than 5 cigarettes per day or average intake of coffee or tea more than 5 cups per day (200 mL/cup) within 3 months before screening, or unable to stop users during the study.
12. With alcohol abuse within 1 year before screening, average weekly alcohol intake more than 14 standard units [1 unit = 360 mL beer (alcohol content 5%) or 45 mL spirits (alcohol content 40%) or 150 mL wine (alcohol content 12%)] or positive for alcohol breath test.
13. With a history of drug abuse within 1 year before screening, or positive for urine drug screening.
14. With a family history of sudden cardiac death (sudden death age less than 40 years).
15. With a resting pulse < 50 beats/min or ≥ 100 beats/min; resting systolic blood pressure < 85 mmHg or ≥ 140 mmHg; resting diastolic blood pressure < 50 mmHg or ≥ 90 mmHg; systolic blood pressure decreased by ≥ 20 mmHg and/or diastolic blood pressure decreased by ≥ 10 mmHg and/or accompanied by clinical symptoms within 3 minutes of standing.
16. Abnormal in 12-lead electrocardiogram (ECG), clinically significant judged by the investigator (e.g., QTcF> 450 ms in men and > 470 ms in women).
17. With the aspartate aminotransferase (AST), alanine aminotransferase (ALT), creatinine (Cr), urea (Urea), serum prolactin levels beyond the upper limit of normal (ULN)，Neutrophil count below the lower limit of normal (LLN).
18. Having special requirements for food, unable to observe a unified diet or having dysphagia.
19. Rejecting abide by the following conditions during the trial: smoking, alcohol or caffeine-containing beverages are prohibited, and strenuous exercise is avoided.
20. Directly related to this clinical trial.
21. Other subjects that the investigator considers inappropriate for this trial.

Adult patients with schizophrenia:

1. Patients who meet the DSM-5 diagnostic criteria for other mental diseases.
2. Patients with refractory schizophrenia to be defined as patients with treatment-resistant schizophrenia who have not achieved clinical improvement after a full course of treatment with at least 2 antipsychotics in the past 5 years.
3. The answer to question 4 or 5 of the Columbia Suicide Scale (C-SSRS) suicide ideation in the screening period is "yes", or the person who has obvious suicide tendency at present or in the past 12 months, or the researcher believes that there is a risk of suicide and violence based on the clinical evaluation of the investigator.
4. There are diseases or functional disorders that affect the clinical trial, including but not limited to neuropsychiatric, cardiovascular, urinary, digestive, respiratory, muscular, metabolic endocrine, hematology, immunology, skin and tumors, etc., clinically significant chronic diseases or poorly controlled diseases that have an impact on this trial as assessed by the investigator.
5. With any surgical condition or condition that may significantly affect the absorption, distribution, metabolism and excretion of the drug, or may pose a hazard to the subjects participating in the trial, such as history of gastrointestinal surgery (gastrectomy, gastrointestinal anastomosis, intestinal resection, etc.), urinary tract obstruction or dysuria, gastroenteritis, gastrointestinal ulcers, history of gastrointestinal bleeding, etc.
6. With a history of epilepsy (except for febrile convulsion).
7. With a history of Malignant syndrome.
8. With a history of severe allergies.
9. Received electric shock treatment, and transcranial magnetic stimulation (rTMS) within 3 months before screening;
10. Subjects are receiving or have recently received (within 5 half-lives, before baseline [Day -1]) oral antipsychotic medications, antidepressants or mood stabilizers.
11. CYP3A4 or CYP2D6 potent inhibitors, moderate inhibitors, potent inducers and moderate inducers used within 5 half-lives before enrollment.
12. Those who have physical examination abnormalities unrelated to schizophrenia at screening, which are judged by the investigator to have an impact on this trial.
13. With a resting pulse < 50 beats/min or ≥ 100 beats/min; resting systolic blood pressure < 85 mmHg or ≥ 140 mmHg; resting diastolic blood pressure < 50 mmHg or ≥ 90 mmHg; systolic blood pressure decreased by ≥ 20 mmHg and/or diastolic blood pressure decreased by ≥ 10 mmHg and/or accompanied by clinical symptoms within 3 minutes of standing.
14. Abnormal in 12-lead electrocardiogram （ECG）, clinically significant judged by the investigator (e.g., QTcF> 450ms in men and > 470ms in women).
15. The laboratory examination during the screening period was abnormal, and the researcher determined that it was of obvious clinical significance, such as: glutamate aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 1.5 times the upper limit of the normal value;creatinine (Cr)>upper limit of normal value;serum prolactin levels ≥ 5 times the upper limit of the normal value
16. With a history of drug abuse within 1 year before screening, or positive for urine drug screening.
17. With alcohol abuse within 1 year before screening, average weekly alcohol intake more than 14 standard units [1 unit = 360mL beer (alcohol content 5%) or 45mL spirits （alcohol content 40%） or 150mL wine （alcohol content 12%）] or positive for alcohol breath test.
18. Rejecting abides by the following conditions during the trial: smoking, alcohol or caffeine-containing beverages are prohibited, and strenuous exercise is avoided.
19. Positive for hepatitis B virus surface antigen （HBsAg）, or syphilis antibody (Anti-TP), or hepatitis C antibody (anti-HCV), or human immunodeficiency virus antigen/antibody combined detection (HIV-Ag/Ab).
20. With a blood donation or blood loss ≥ 400mL within 3 months before screening, or a blood donation or blood loss ≥ 200mL within 1 month.
21. Participation in another clinical study within 3 months before screening in which the subject received an experimental or investigational drug agent,or are participating in clinical trials.
22. Other subjects that the investigator considers inappropriate for this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-16 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Baseline to 15 days after the last administration
  Incidence of Treatment-Emergent Adverse Events

SECONDARY OUTCOMES:
Cmax | Baseline to 360 hours after the last administration
  maximum observed plasma concentration of VV119 and the main metabolites
area under the plasma concentration time curve from time zero to the last (AUC0-t) | Baseline to 360 hours after the last administration
  area under the plasma concentration time curve from time zero to the last of VV119 and the main metabolites
AUC0-∞ | Baseline to 360 hours after the last administration
  area under the plasma concentration time curve from time zero to infinity of VV119 and the main metabolites
Tmax | Baseline to 360 hours after the last administration
  time at which Cmax occurs of VV119 and the main metabolites of VV119 and the main metabolites
t1/2 | Baseline to 360 hours after the last administration
  half-life of elimination of VV119 and the main metabolites
Apparent Clearance Rate（CL/F） | Baseline to 360 hours after the last administration
  apparent clearance of VV119 and the main metabolites
Vd/F | Baseline to 360 hours after the last administration
  apparent volume of distribution during the terminal phase of VV119 and the main metabolites
Ke | Baseline to 360 hours after the last administration
  elimination rate constant of VV119 and the main metabolites
AUC0-24h | Baseline to 360 hours after the last administration
  area under the plasma concentration time curve from time zero to 24h of VV119 and the main metabolites
mean Resident Time | Baseline to 360 hours after the last administration
  mean Resident Time from time zero to infinity/the last of VV119 and the main metabolites
Positive and Negative Syndrome Scale （PANSS） | Day-1,Day14,Day28 and Day42
  Change from Baseline in Positive and Negative Syndrome Scale in part Ⅱ。 The PANSS measures symptom severity of participants with schizophrenia and contains 7 positive symptom scales,7negative system scales, and 16 general psychopathology symptom scales. Participants are rated from 1 to 7 on each symptom scale with a total minimum score of 30 and a maximum score of 210. A decrease in PANSS total score correlates with an improvement in schizophrenia symptoms.
PANSS Positive subscale score | Day-1, Day14, Day28 and Day42
  Change from Baseline in PANSS Positive subscale score in part Ⅱ PANSS-Positive: Assessment of positive symptoms. Minimum value:7, maximum value:49, the higher scores mean a worse outcome.
PANSS Negative subscale score | Day-1, Day14, Day28 and Day42
  Change from Baseline in PANSS Negative subscale score in part Ⅱ。 PANSS-negative: Assessment of negative symptoms. Minimum value:7, maximum value:49, the higher scores mean a worse outcome.
Treatment response rate | Day-1,Day14, Day28 and Day42
  Positive and Negative Syndrome Scale （PANSS） Response rate, Defined as a 50% or Greater Improvement from Baseline in PANSS Total Score in part Ⅱ
Clinical Global Impression-Severity (CGI-S) | Day-14, Day28 and Day42
  Change from Baseline in Clinical Global Impression-Severity in part Ⅱ。 The CGI-S rating scale is a 7-point global assessment that measures the clinician's impression of the severity of illness exhibited by a participant. A rating of 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill participants". Negative change from baseline scores indicate improvement in the severity of illness.
Rac | Baseline to 360 hours after the last administration
  Accumulation Ratio of VV119

CONTACTS AND LOCATIONS:
Overall Officials: Gang Wang, Principal Investigator — Beijing Anding Hospital of Capital Medical University
Locations (3):
- China (3):
  - Beijing Anding Hospital of Capital Medical University, Beijing, Beijing Municipality
  - Beijing Huilongguan Hospital, Beijing, Beijing Municipality
  - Xi'an Mental Health Center, Xi’an, Shanxi

IPD SHARING:
Plan to Share IPD: No